CLINICAL TRIAL: NCT00238550
Title: Randomised Control Trial Studying the Addition of CBME to Conventional Treatment for the Relief of Painful Diabetic Neuropathy
Brief Title: Study of CBME in the Relief of Painful Diabetic Neuropathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Collaborators: Diabetes UK (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STH9042 02/343; BDA:RD03/0002590
Record Dates: First submitted 2005-10-12; First posted 2005-10-13 (Estimated); Last update posted 2022-06-13 (Actual); Status verified 2022-06

CONDITIONS: Diabetic Neuropathy; Painful
Keywords: Diabetes; Pain; Peripheral neuropathy
MeSH Terms: conditions — Diabetic Neuropathies; Pain; Diabetes Mellitus; Peripheral Nervous System Diseases

INTERVENTIONS:
Drug: Cannabis based medicine extract (CBME)

SUMMARY:
The study is designed to investigate the benefit of adding CBME to the existing treatment regime in the management of painful neuropathy.

Hypothesis:

1. The addition of CBME to the existing treatment regime will result in a significant improvement in both primary and secondary outcome measures.
2. The side effect profile and tolerability of CBME will be minimal and comparable to placebo.

DETAILED DESCRIPTION:
1. To investigate the benefit of adding CBME to the existing treatment regime in the management of painful neuropathy.
2. To study the tolerability and side effect profile of CBME.
3. To study the effects of CBME treatment on vibration perception thresholds (VPT) and nerve conduction study parameters.
4. To evaluate the effects of CBME on central nervous system deep nuclei using MR Spectroscopy.

ELIGIBILITY:
Inclusion Criteria:

Diagnoses of diabetes will be based on the criteria set by the World Health Organisation.

Subjects must be over 18 years of age. Female subjects of child bearing potential and male subjects whose partner is of child bearing potential must be willing to ensure that they or their partner use effective contraception during the study and for three months thereafter.

Written consent will be obtained. Volunteers must have had symptoms consistent with painful neuropathy for at least six months to be eligible for recruitment (NTSS 6 score of greater than 4 and less than 16).

Subjects in whom the symptoms of painful neuropathy persist despite an adequate trial with tricyclic antidepressants (TCA).

Stable dose of current treatment for neuropathy for at least 3 months prior to entry into the study.

Able (in the investigators opinion) and willing to comply with all study requirements.

Willing to allow his or her GP and consultant, if appropriate, to be notified of participation in the study.

Willing to allow his or her name to be notified to the Home Office and GW Pharma for participation in this study.

Exclusion Criteria:

Previous cerebrovascular events or other neurological disorders. unstable glycaemic control for six months. History of cardiovascular disorders. History of schizophrenia or any other psychiatric illnesses other than depression associated with painful diabetic neuropathy History of epilepsy. Serious illnesses precluding the gathering of or potentially having an impact on primary and secondary outcome measures for example major organ failure, neoplasia or coeliac disease.

Unwilling to stop driving or operating dangerous machinery for four hours after dosing on study medication or if experiencing its side effects.

Anticipated foreign travel within the first 15 weeks of the trial. Participants in other research studies currently or within the previous three months.

Current or past history of substance abuse. Previous or current history of consuming more than 20 units of alcohol a week. Neuropathy due to other aetiologies. Known or suspected hypersensitivity to cannabinoids or any of the excipients of the study medications.

Known or suspected adverse reaction to cannabinoids. Pregnancy or lactating mothers or planning pregnancy during the course of the study.

Not using adequate contraception Current use of fentanyl Significant renal or hepatic impairment as shown in medical history or indicated by clinical laboratory results from samples taken at baseline.

Scheduled elective surgery or other procedures requiring general anaesthesia during the study.

Regular levodopa therapy within 7 days of study entry. Severe cognitive impairment such that the patient is unable to provide informed consent.

Donation of blood during the study Other problems likely to make participation difficult at the discretion of the Treatment Physician

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2003-10; Study Completion 2006-03

PRIMARY OUTCOMES:
Improvement in pain symptoms, including pain perception and sleep quality, utilising daily diaries and validated pain questionnaires during 12 week treatment period and after 3 month cessation of treatment

SECONDARY OUTCOMES:
1.Quality of life utilising validated questionnaires
questionnaires.
2.Evaluation of the tolerability and side effect profile of the study medication will be employed.
3. Neurophysiology including assessment of sensory and motor nerve function to the lower limbs.
(1, 2 & 3: During the 12 week treatment period and after 3 month cessation of treatment)
4. Magnetic Resonance Imaging
MR spectroscopy of the chemical constituents in the deep nuclei of the brain will be analysed before and after 12 week treatment period.

CONTACTS AND LOCATIONS:
Overall Officials: Solomon Tesfaye, Principal Investigator — Sheffield Teaching Hosiptals NHS Foundation Trust
Locations (1):
- Royal Hallamshire Hospital, Sheffield, South Yorkshire, United Kingdom